CLINICAL TRIAL: NCT05907798
Title: Effect of Serratus Anterior Plan Block (SAP) and Pectoralis (PECSI-II) Peripheral Blocks on Left Internal Mammarian Artery (LIMA) Blood Flow in Coronary Bypass Surgery
Brief Title: Serratus Anterior Plan Block (SAP) and Pectoralis (PECSI-II) Blocks on Left Internal Mammarian Artery (LIMA) Blood Flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Arzu Esen Tekeli, Associate Professor, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2023-4
Record Dates: First submitted 2023-05-23; First posted 2023-06-18 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Chest Wall Blocks

STUDY DESIGN:
Intervention Model Description: Randomized, single-blind, method comparison study
Who Masked: Participant
Masking Description: Patients will be randomly divided into 3 groups using the closed envelope method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group PECS (Active Comparator): placing the ultrasound probe in the midclavicular line and in the parasagittal plane, After identifying the second and third ribs by sliding the ultrasound probe caudally, the lower end will be rotated towards the axilla to make the probe parallel to the deltopectoral groove. Combined with the in-plane technique, this rotation provides better extension to the intercostobrachial nerve. The tip of the needle will be inserted into the interpectoral fascial plane (between pectoralis major and minor). The needle will be advanced from the interpectoral fascial plane to the fascial plane between the pectoralis minor and the serratus anterior. 10 mL of local anesthetic (Bupivacaine) will be applied to the PECS I area and 20 mL to the PECS II area.
  Interventions: Procedure: LIMA Blood flow
- Group SA (Active Comparator): It will be positioned to stand at the head of the patient or to one side of the patient and to see the ultrasound screen easily. High-frequency linear probe and 80 mm blunt-tipped needle will be placed cauda-cranially or cranially-caudal with in-plane technique. The injection site is found by placing the ultrasound probe under the clavicle in a parasagittal manner and counting from the second rib. By moving the probe laterally towards the mid or posterior axillary line, the serratus anterior muscle is seen as a layer of muscle over the anechoic shadow of the rib. It extends over the latissimus dorsi serratus anterior muscle and appears thicker and more prominent in the posterior axillary line. 30 mL of local anesthetic (bupivacaine) will be administered to the fascial plane by advancing the needle superficially or deeply into the serratus anterior muscle.
  Interventions: Procedure: LIMA Blood flow
- Group K (Control group) (Sham Comparator): The patient, who was taken to the operating table with his consent, will be monitored. ECG monitoring, SpO2 monitoring, invasive artery monitoring will be performed. General Anesthesia will be applied(Induction with 2 mg/kg propofol, 0.6mg/kg rocuronium bromide, 2µcg/kg fentanyl, 2MAC sevoflurane + 40% air mixture and maintenance with 2L/min) Routine coronary artery bypass grafting surgery will be performed without any peripheral blocking and LIMA blood flow will be measured.
  Interventions: Procedure: LIMA Blood flow

INTERVENTIONS:
Procedure: LIMA Blood flow — 30 minutes after induction

SUMMARY:
To investigate whether the anterior chest wall blocks performed before the surgery have an effect on the LIMA (left internal mammarian artery) blood flow in patients who will undergo coronary artery bypass surgery.

DETAILED DESCRIPTION:
Coronary artery bypass grafting (CABG), also known as heart bypass surgery, is a procedure performed to improve reduced blood flow due to narrowing of the coronary arteries. The left internal mammary artery (LIMA) is generally the preferred perforator artery for grafting of the left anterior descending (LAD) coronary artery from the coronary arteries. However, spasm during the release phase for anastomosis often complicates surgical dissection and anastomosis, and adversely affects flow dynamics (1) LIMA has been used as an important potential graft in coronary artery bypass graft (CABG) surgery since the 1970s. LIMA has a potent biological function through the production of vasodilator and platelet inhibitory factors. LIMA's feature of having less fenestration, lower intimal hyperplasia tendency and less permeability in intercellular connections prevents lipoproteins from entering the subendothelial space (2) The use of ultrasound in anesthesia practice, especially for analgesia, is increasingly popular. The sonoanatomical dominance of anesthetists on regional structures is increasing, especially with plan blocks, a new one being defined every day. The primary aim of this study was to investigate the effect of the ultrasound guided papaverine application method and the traditional method of topical papaverine application on the LIMA flow measured before and after anastomosis. Papaverine will be administered to all patients after the block procedure at the beginning of the surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* Agreeing to participate in the study
* 20-65 years old
* ASA I-II-III
* Coronary artery bypass grafting will be performed

Exclusion Criteria:

* Refusal to participate in the study
* Patients under the age of 20, over the age of 65
* presence of pregnancy
* Bleeding diathesis
* Liver or kidney failure
* Acute and bleeding patients Those who receive inotropic support starting from the preoperative period
* BMI ≥30

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2024-06-02 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Blood flow | 30 minutes after induction
  LIMA blood flow will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Medicine School Department of Anesthesiology and Reanimation, Study Chair — Yuzuncu Yil University
Locations (1):
- Arzu Esen Tekeli, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Participants' personal information will not be shared.